CLINICAL TRIAL: NCT00965107
Title: Onset Time of Thiopental Versus Propofol in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Lars Rasmussen, Department of Anesthesia, Center of Head and Orthopedics, Copenhagen University Hospital Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1A-AGE/ONSET
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-02

CONDITIONS: Induction of Anaesthesia; Age
MeSH Terms: interventions — Thiopental; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thiopental (Experimental): Thiopental for induction of anaesthesia.
  Interventions: Drug: Thiopental
- Propofol (Active Comparator): Propofol for induction of anaesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Thiopental — Thiopental given as a bolus dose of 2,5 mg/kg.
  Other Names: Thiomebumalnatrium, thiomebumal
  Arms: Thiopental
Drug: Propofol — Propofol given as a bolus dose of 1 mg/kg.
  Arms: Propofol

SUMMARY:
This study is aimed at increasing the safety of the use of anaesthesia in an elderly population (> 60 years). Patients with decreased physiological reserve, including all elderly patients, have an increased risk of getting an erroneous induction bolus. This project will investigate how fast elderly patients (> 60 years) fall asleep during bolus induction of anaesthesia with two of the most used hypnotics, thiopental and propofol, evaluated with BIS-monitoring and clinical signs of anaesthetic depth. The hemodynamic response will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients above 60 years of age, with an indication of general anaesthesia during surgery.
* Informed consent.
* The patient must be legally competent.
* The patient must be able to read and understand Danish.

Exclusion Criteria:

* Known allergic reactions to thiopental, propofol, lidocaine or alfentanil
* "Body Mass Index" (BMI) <18 and > 35.
* NYHA-class > 2.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
"Onset-time" defined as the time from started induction bolus to: - Time to BIS-value <50. | 120 seconds

SECONDARY OUTCOMES:
Hemodynamical effect (bloodpressure/pulse) every 60 seconds. | 120 seconds
"Onset-time" defined as the time from started induction bolus to: - Time to loss of grip. | 120 seconds
"Onset-time" defined as the time from started induction bolus to: - Time to eye closure. | 120 seconds
"Onset-time" defined as the time from started induction bolus to: - Time to ciliary reflex cessation. | 120 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rasmussen, MD, PHD, Principal Investigator — Rigshospitalet, Denmark; Martin K Soerensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Anesthesia, Center of Head and Orthopedics, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Department of Anesthesia, Juliane Marie Center, Copenhagen University Hospital Rigshospitalet, Copenhagen